CLINICAL TRIAL: NCT06083766
Title: Metabolic and Physiologic Responses to Hormone Therapy in Transgender and Gender Diverse People
Status: Recruiting | Type: Observational
Sponsor: Mayo Clinic (Other)
Responsible Party: Principal Investigator, K. Sreekumaran Nair, Principal Investigator, Mayo Clinic
Other Study IDs: 23-006826
Record Dates: First submitted 2023-10-09; First posted 2023-10-16 (Actual); Last update posted 2025-11-10 (Actual); Status verified 2025-11

CONDITIONS: Effects of GAHT, on Skeletal Muscle in TGD
Keywords: Transgender; Gender Diverse

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Biospecimen Retention: Samples With DNA — whole blood, serum, white cells, urine, tissue
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Transmasculine/transfeminine individuals and/or transgender men/women (whom are NOT receiving GAHT)
  Interventions: Behavioral: hormone therapy
- Transmasculine/transfeminine individuals and/or transgender men/women (whom ARE receiving GAHT)
  Interventions: Behavioral: hormone therapy

INTERVENTIONS:
Behavioral: hormone therapy — Determine how gender affirming hormone therapy affects muscle physiology

SUMMARY:
The primary purpose of this research is to determine how gender affirming hormone therapy affects muscle physiology.

DETAILED DESCRIPTION:
Study participation involves a screening visit and two study visits. The screen includes blood draws, and urine testing. The first visit requires a collection of breath, exercise testing, and body scans. Between visits participant are to eat three days of provided meals and wear an activity monitor. The second study visit will be 3-14 days after the first and includes blood draws, a meal test, and a muscle biopsy. If individuals are not on gender affirming hormone therapy at the time of participation, they may be able to participate again if you decide to pursue gender affirming hormone therapy later on.

ELIGIBILITY:
Inclusion Criteria:

* age 18-40yrs
* BMI 18.5-38 kg/m2
* Fasting glucose < 100 mg/dL
* No gender affirming gonadal surgery

We seek to enroll 6 patients in each group who have been on GAHT for more than 10 months with minimal interruptions in treatment.

Exclusion Criteria:

* Pregnancy
* Use of hormonal forms of birth control within the previous 3 months
* Use of glucocorticoids, estradiol, testosterone, progestin, antiandrogens, or antiestrogens besides those received as part of a supervised hormone therapy.
* Gender-affirming gonadal surgery
* Prior use of gonadotropin releasing hormone (GnRH) analogues during puberty
* Coronary artery disease or heart failure.
* A known medical condition that in the judgment of the investigator might interfere with the completion of the protocol such as the following examples:

  * Inpatient psychiatric treatment in the past 6 months
  * Presence of a known adrenal disorder
  * Abnormal liver function test results (Transaminase >2 times the upper limit of normal); testing required for subjects taking medications known to affect liver function or with diseases known to affect liver function
  * Abnormal renal function test results (calculated GFR <45 mL/min/1.73m2); testing required for subjects with diabetes duration of greater than 5 years post onset of puberty
  * Active gastroparesis
  * If on antihypertensive, thyroid, anti-depressant or lipid lowering medication, lack of stability on the medication for the past 2 months prior to enrollment in the study
  * Uncontrolled thyroid disease (TSH undetectable or >10 mlU/L); testing required within three months prior to admission for subjects with a goiter, positive antibodies, or who are on thyroid hormone replacement, and within one year otherwise
  * Abuse of alcohol or recreational drugs
  * Infectious process not anticipated to resolve prior to study procedures (e.g. meningitis, pneumonia, osteomyelitis).
  * Uncontrolled arterial hypertension (Resting diastolic blood pressure >90 mmHg and/or systolic blood pressure >160 mmHg) at the time of screening.
  * A recent injury to body or limb, muscular disorder, use of any medication, any carcinogenic disease, or other significant medical disorder if that injury, medication, or disease in the judgment of the investigator will affect the completion of the protocol (exercise testing or muscle biopsy).
  * Medications that may impact study end points such as mitochondrial biology e.g. beta blockers
  * Anti-hyperglycemic drugs including metformin
  * Any other medication that the investigator believes is a contraindication to the subject's participation.

Ages: 18 Years to 40 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: Transgender and Gender Diverse People Residents within a 100-mile radius of Mayo Clinic, Rochester, MN.
Sampling Method: Non-Probability Sample
Enrollment: 24 (Estimated)
Dates: Start 2024-01-04 (Actual); Primary Completion 2026-04 (Estimated); Study Completion 2026-07 (Estimated)

PRIMARY OUTCOMES:
Aim 1 | 2 weeks
  To identify the impact of gender-affirming hormone therapy (GAHT) on skeletal muscle mitochondrial metabolism in transgender and gender diverse individuals.

SECONDARY OUTCOMES:
Aim 2 | 2 weeks
  To determine changes in important parameters of physiologic and functional health following gender-affirming hormone therapy (GAHT) in and gender diverse people.

CONTACTS AND LOCATIONS:
Locations (1):
- Mayo Clinic, Rochester, Minnesota, United States

IPD SHARING:
Plan to Share IPD: Undecided